CLINICAL TRIAL: NCT03294369
Title: RIesgo CARdiovascular y Eventos Cardiovasculares en la población General Del área Sanitaria de TOledo
Brief Title: Cardiovascular Risk in Toledo Population
Acronym: RICARTO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Castilla-La Mancha Health Service (Other)
Collaborators: Castile-La Mancha Government (Socio-Sanitary Foundation of Castile-La Mancha) (Unknown); SEMERGEN (Spanish Society of Primary Care Physicians) (Unknown)
Responsible Party: Principal Investigator, Gustavo Rodriguez Roca, Director & principal Investigator, Clinical Professor, Castilla-La Mancha Health Service
Other Study IDs: RICARTO
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Cardiovascular Risk Factor; Cardiovascular Diseases
Keywords: Hypertension; Diabetes; Dyslipidemia; Smoking; Cardiovascular; Toledo
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Diabetes Mellitus; Dyslipidemias; Smoking | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Total blood and serum samples will be frozen (-85ºC) for future genetic studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of the study: A sample from the general population aged 18 years or older, randomly selected from a database of sanitary cards stratified by age and gender.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This is an observational study. No specific diagnostic or therapeutic procedure will be performed due to the study.

SUMMARY:
This epidemiological and observational study is aimed to assess cardiovascular risk (CVR) by investigating the prevalence of CVR factors (CVRF), target organ damage (TOD) and cardiovascular disease (CVD) in general population of the sanitary area of Toledo.

DETAILED DESCRIPTION:
Epidemiological and observational study that is analyzing a sample from the general population aged 18 years or older, randomly selected from a database of sanitary cards stratified by age and gender.

Clinical history, physical examination and complementary tests are being performed.

Total blood and serum samples are being frozen (-85ºC) for future genetic studies. The biobank is currently being registered at the "Virgen de la Salud" hospital of Toledo.

CVR is assessed by SCORE scale calibrated for Spanish population and the Framingham Heart Study scale.

Patients will be periodically visited, with a minimum follow-up of 5 years. Standard statistical analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or older, randomly selected from a database of health cards stratified by age and gender

Exclusion Criteria:

* Individulas aged under 18 years.
* Subjects who do not sign the informed consent.
* Subjects that due to different conditions (physical, mental or social) is expected that do not complete the expected follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged 18 years or older, randomly selected from a database of health cards stratified by age and gender
Sampling Method: Probability Sample
Enrollment: 3125 (Estimated)
Dates: Start 2011-04-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess cardiovascular risk of the study population | December 2020
  Cardiovascular risk will be determined according to SCORE scale calibrated for Spanish population and the Framingham Heart Study scale.
Prevalence of cardiovascular risk factors | December 2020
  To assess the prevalence of cardiovascular risk factors
Prevalence of cardiovascular disease | December 2020
  To assess the prevalence of cardiovascular disease

CONTACTS AND LOCATIONS:
Locations (1):
- Avenida de Irlanda, 12, 2º A, Toledo, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rodriguez-Roca GC, Segura-Fragoso A, Villarin-Castro A, Alonso-Moreno FJ, Rodriguez-Padial L, Rodriguez-Garcia ML, Fernandez-Conde JA, Rojas-Martelo GA, Menchen-Herreros A, Escobar-Cervantes C, Fernandez-Martin J, Artigao-Rodenas LM, Carbayo-Herencia JA, Hernandez-Moreno J; en representacion del grupo de trabajo RICARTO. [Characteristics and cardiovascular events in a general population included in the RICARTO (RIesgo CARdiovascular TOledo) study: Data from the first 1,500 individuals included in the study]. Semergen. 2018 Apr;44(3):180-191. doi: 10.1016/j.semerg.2017.07.002. Epub 2017 Aug 30. Spanish. PMID 28869129
- [Result] Rodriguez-Roca GC, Rodriguez-Padial L, Alonso-Moreno FJ, Segura-Fragoso A, Villarin-Castro A, Rodriguez-Garcia ML, Menchen-Herreros A, Rojas-Martelo GA, Fernandez-Conde JA, Artigao-Rodenas LM, Carbayo-Herencia JA, Escobar-Cervantes C, Hernandez-Moreno J, Fernandez-Martin J; en representacion del grupo de trabajo RICARTO. [Cardiovascular risk and cardiovascular events in the general population of the sanitary area of Toledo. RICARTO Study]. Semergen. 2018 Mar;44(2):107-113. doi: 10.1016/j.semerg.2017.04.007. Epub 2017 May 27. Spanish. PMID 28566229
- [Result] Rodriguez-Roca GC, Villarin-Castro A, Carrasco-Flores J, Artigao-Rodenas LM, Carbayo-Herencia JA, Escobar-Cervantes C, Alonso-Moreno FJ, Segura-Fragoso A, Gomez-Serranillos M, Hernandez-Moreno J; RICARTO (Riesgo Cardiovascular Y Eventos Cardiovasculares En La Poblacion General del Area Sanitaria De Toledo) Project Working Group. Concordance between automated oscillometric measurement of ankle-brachial index and traditional measurement by eco-Doppler in patients without peripheral artery disease. Blood Press. 2014 Oct;23(5):270-5. doi: 10.3109/08037051.2013.876796. Epub 2014 Mar 19. PMID 24646328
- [Result] Rodriguez-Roca GC, Rodriguez-Padial L, Alonso-Moreno FJ, Romero-Gutierrez A, Akerstrom F, Segura-Fragoso A, Villarin-Castro A, Hernandez-Moreno J, Menchen-Herreros A, Gomez-Serranillos M, Artigao-Rodenas LM; grupo de trabajo del estudio RICARTO. [Lipid profile in patients admitted with acute coronary syndrome in Spain: data from Toledo health care area between 2005 and 2008]. Semergen. 2013 Sep;39(6):298-303. doi: 10.1016/j.semerg.2012.11.001. Epub 2012 Dec 20. Spanish. PMID 24034757
- [Result] Rodriguez Padial L, Segura Fragoso A, Alonso Moreno FJ, Arias MA, Villarin Castro A, Rodriguez Roca GC. Blood pressure differences between one automatic measurement and the mean value of 3 automatic measurements. SPRINT trial. Med Clin (Barc). 2017 Jul 21;149(2):72-74. doi: 10.1016/j.medcli.2017.01.013. Epub 2017 Mar 9. English, Spanish. PMID 28284813